CLINICAL TRIAL: NCT01141712
Title: High Dose Chemotherapy With Autologous Stem Cell Rescue for Aggressive B Cell Lymphoma and Hodgkin Lymphoma in HIV-infected Patients (BMT CTN #0803)
Brief Title: Autologous Transplant in HIV Patients (BMT CTN 0803)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0803; U01HL069294 (NIH); U01HL069294-06 (NIH); U01CA121947 (NIH)
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Lymphoma; HIV
Keywords: HIV; B-cell Lymphoma; Burkitt's Lymphoma; Follicular Lymphoma; Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma, Follicular; Hodgkin Disease | interventions — Transplantation, Autologous; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous transplant (Other): Patients will receive BCNU 300 mg/m^2 Day -6, Etoposide 100 mg/m^2 BID Days -5 to -2, Cytarabine 100 mg/m^2 BID Days -5 to -2, and Melphalan 140 mg/m^2 Day -1 followed by autologous HCT.
  Interventions: Procedure: Autologous transplant; Drug: BCNU; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan

INTERVENTIONS:
Procedure: Autologous transplant — Participants will receive the BEAM conditioning regimen followed by autologous HCT.
Drug: BCNU — Participants will receive BCNU 300 mg/m^2 Day -6
  Other Names: Carmustine
Drug: Etoposide — Participants will receive Etoposide 100 mg/m^2 BID Days -5 to -2
  Other Names: VP-16
Drug: Cytarabine — Participants will receive Cytarabine 100 mg/m^2 BID Days -5 to -2
  Other Names: Depocyt
Drug: Melphalan — Participants will receive Melphalan 140 mg/m^2 Day -1
  Other Names: Alkeran

SUMMARY:
This study is a Phase II, multicenter trial assessing overall survival after autologous hematopoietic stem cell transplantation using a BEAM transplant regimen (carmustine, etoposide, cytarabine, melphalan) in lymphoma patients with HIV.

DETAILED DESCRIPTION:
BACKGROUND:

Non-Hodgkin lymphoma (NHL) is an AIDS-defining diagnosis for patients infected with the Human Immunodeficiency Virus (HIV). While the incidence of NHL has decreased amongst HIV-infected patients since the advent of highly-active anti-retroviral therapy (HAART), lymphoma remains a significant cause of death for this patient population. The prognosis for patients with AIDS-related lymphoma is dramatically different in the era of HAART therapy. In a comparison of treatment outcomes for patients treated before and after the advent of HAART, there is a statistically significant improvement in the overall survival of patients treated with HAART. Unfortunately, despite considerable advances in the treatment of AIDS-related NHL, induction-failure and disease relapse remain key challenges. The prognosis for patients with refractory and relapsed NHL is poor with overall survival rates of less than 20 percent for patients treated with non-transplant salvage therapies. Based upon a randomized trial and numerous phase II trials, high-dose therapy with autologous hematopoietic cell transplantation (HCT) has been established as the standard of care for patients with chemotherapy-sensitive relapsed non-Hodgkin lymphoma.

DESIGN NARRATIVE:

All patients must have chemosensitive disease as demonstrated by response to induction or salvage chemotherapy. Patients must also have less than or equal to 10percent bone marrow involvement after their most recent salvage therapy. Patients cannot have had prior autologous or allogeneic HCT. Patients must initiate conditioning therapy within 3 months of mobilization or bone marrow harvest.

Mobilization therapy may be employed per institutional guidelines. Patients must have an adequate autograft to be eligible for the protocol. Patients may not have HIV refractory to pharmacologic therapy. Patients must not have opportunistic infection that is not responding to therapy. Patients will receive Carmustine (BCNU) 300 mg/m^2 Day -6, Etoposide 100 mg/m^2 twice a day (BID) on Days -5 to -2, Cytarabine 100 mg/m2 BID on Days -5 to -2, and Melphalan 140 mg/m2 Day -1 followed by autologous HCT.

Patients will be followed for 2 years post-transplant. Survival data, time to progression data, progression-free survival data, time to progression after Complete Remission (CR) data, lymphoma disease-free survival data, time to hematopoietic recovery data, hematologic function data, toxicity data, incidence of infections, treatment-related mortality data, immunologic reconstitution data, data assessing the impact of therapy on the HIV reservoir and microbial gut translocation will be recorded and reported periodically to the BMT CTN Data and Coordinating Center (DCC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of persistent or recurrent World Health Organization (WHO) classification diffuse large B-cell lymphoma, composite lymphoma with > 50% diffuse large B-cell lymphoma, mediastinal B-cell lymphoma, immunoblastic, plasmablastic, Burkitt's or Burkitt-like or classical Hodgkin's lymphoma. Patients transformed from follicular lymphoma are eligible for the study, pending fulfillment of other criteria.
* 15 years old or older
* Three or fewer prior regimens of chemotherapy over the entire course of their disease treatment (including one induction chemotherapy and no more than 2 salvage chemotherapies). Monoclonal antibody therapy and involved field radiation therapy will not be counted as prior therapies.
* All patients must have chemosensitive disease as demonstrated by at least a partial response to induction or salvage therapy.
* Less than or equal to 10% bone marrow involvement.
* Patients with adequate organ function as measured by: a)Cardiac: American Heart Association Class I: Patients with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain. Additionally, all patients must have a left ventricular ejection fraction at rest greater than or equal to 40% demonstrated by Multi Gated Acquisition Scan (MUGA) or echocardiogram; b)Hepatic: (i) Bilirubin less than 2.0 mg/dL (except for isolated hyperbilirubinemia attributed to Gilbert syndrome or antiretroviral therapy) and alanine transaminase (ALT) and aspartate transaminase (AST) greater than 3x the upper limit of normal; (ii) Concomitant Hepatitis: Patients with chronic hepatitis B or C may be enrolled on the trial providing the above criteria are met. In addition, no active viral replication - undetectable (viral load less than 500 copies/ml) hepatitis B DNA level by PCR and no clinical or pathologic evidence of irreversible chronic liver disease; c)Renal: Creatinine clearance (calculated creatinine clearance is permitted) greater than 40 mL/min; d)Pulmonary: Carbon Monoxide Diffusing Capacity (DLCO), forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) greater than or equal to 45% of predicted (corrected for hemoglobin).
* Autologous peripheral stem cell graft with a minimum of greater than or less than 1.5 x 10^6 CD 34+ cells/kg (target greater than or less than 2.0 x 10^6 CD 34+ cells/kg) or if peripheral blood stem cell (PBSC) mobilization fails, cells can be obtained by bone marrow harvest per institutional practices (in cases where bone marrow will be used for transplantation, the required CD34+ dose does not apply and institutional requirements for total nucleated cell dose should apply).
* Initiate conditioning therapy within 3 months of mobilization or bone marrow harvest.
* Signed informed consent.
* Patients on antiretroviral therapies (ARVs) can either have: a) Undetectable HIV viral load (VL less than 50 copies); b) If VL detectable at less than 2000 copies/mL must have review of previous antiretroviral regimens or previous genotypic or phenotypic testing which indicate the ability to fully suppress virus by addition of sensitive drugs. This review will be carried out by the Infectious Disease (ID) specialist caring for the patient; c)If VL detectable at greater than 2000 copies/mL, a current HIV genotype and/or phenotype must be obtained. If a HAART regimen to which the patient's virus is sensitive can be determined based on genotype and previous antiretroviral experience, then the patient will be considered eligible in this regard. This review will be carried out by the ID specialist caring for the patient.

Exclusion Criteria:

* Karnofsky performance score less than 70%.
* Uncontrolled bacterial, viral or fungal infection (currently taking medication and with progression or no clinical improvement).
* Prior malignancy in the 5 years prior to enrollment except resected basal cell carcinoma, treated cervical carcinoma in situ or Kaposi's sarcoma: a)Symptomatic Kaposi's sarcoma currently requiring therapy is excluded (patients receiving topical therapy for minimal disease are not included in this definition); b)Prior treatment with topical agents, local radiation, or up to 6 cycles of cytotoxic chemotherapy at least six months prior is permitted; c) Other cancers treated with curative intent less than 5 years previously will not be allowed unless approved by the Medical Monitor or Protocol Chair; d)Cancer treated with curative intent more than 5 years previously will be allowed.
* Pregnant (positive β-HCG) or breastfeeding.
* Fertile men or women unwilling to use contraceptive techniques from the time of initiation of mobilization until six-months post-transplant.
* Prior autologous or allogeneic HCT.
* Patients with evidence of Myelodysplastic Syndrome (MDS)/Acute Myeloid Leukemia (AML) or abnormal cytogenetic analysis indicative of MDS on the pre-transplant bone marrow examination. Pathology report documentation need not be submitted.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-04; Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (16):
- United States (16):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego Medical Center, La Jolla, California
  - UCLA, Los Angeles, California
  - University of CA, SF, San Francisco, California
  - University of Florida College of Medicine, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - BMT Program at Northside Hospital, Atlanta, Georgia
  - University of Maryland Medical Systems, Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins Medical Institution, Baltimore, Maryland
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Texas/MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Alvarnas JC, Le Rademacher J, Wang Y, Little RF, Akpek G, Ayala E, Devine S, Baiocchi R, Lozanski G, Kaplan L, Noy A, Popat U, Hsu J, Morris LE Jr, Thompson J, Horowitz MM, Mendizabal A, Levine A, Krishnan A, Forman SJ, Navarro WH, Ambinder R. Autologous hematopoietic cell transplantation for HIV-related lymphoma: results of the BMT CTN 0803/AMC 071 trial. Blood. 2016 Aug 25;128(8):1050-8. doi: 10.1182/blood-2015-08-664706. Epub 2016 Jun 13. PMID 27297790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between April 2010 and March 2013 from 16 different transplant centers.
Pre-assignment Details: Three patients did not undergo transplantation due to disease progression prior to conditioning.
Groups:
- Autologous Transplant: Patients will receive BCNU 300 mg/m^2 Day -6, Etoposide 100 mg/m^2 twice a day from Days -5 to -2, Cytarabine 100 mg/m^2 twice a day from Days -5 to -2, and Melphalan 140 mg/m^2 Day -1 followed by autologous HCT.
Period: Overall Study
Arm/Group | Autologous Transplant
Started | 43
Completed | 40
Not Completed | 3
Not completed — Disease progression | 3

BASELINE CHARACTERISTICS:
Groups:
- Autologous Transplant: Patients will receive BCNU 300 mg/m^2 Day -6, Etoposide 100 mg/m^2 twice a day (BID) on Days -5 to -2, Cytarabine 100 mg/m^2 BID Days -5 to -2, and Melphalan 140 mg/m^2 Day -1 followed by autologous HCT.
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 46.9 [22.5 to 62.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 13
  White | 24
  Unknown | 3
Karnofsky Performance Score [Number; unit: participants] — Measure Description: Assesses patient self-perceived global quality of life and functioning on a scale of 0 - 100; where 100 equals normal quality of life with no evidence of disease, 90 equals ability to carry on normal activity with minor signs/symptoms of disease, 80 equals normal activity with effort and some signs/symptoms of disease, and 70 equals ability to care for self but unable to carry on normal activity or to do active work.
  participants
    100 | 11
    90 | 20
    80 | 7
    70 | 2
Participant Diagnosis [Number; unit: participants]
  Hodgkin's Lymphoma | 15
  Diffuse Large B-cell Lymphoma | 16
  Plasmablastic Lymphoma | 2
  Burkitt's Lymphoma | 7
Disease Status [Number; unit: participants]
  Complete Remission | 30
  Partial Remission | 9
  Relapsed or Progressive Disease | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Assess the OS after autologous hematopoietic stem cell transplantation (HCT) for chemotherapy-sensitive aggressive B cell lymphoma or Hodgkin's lymphoma in patients with HIV using BEAM for pre-transplant conditioning. The primary analysis will consist of estimating the 1 year OS probability from the time of transplantation based on the Kaplan-Meier product limit estimator. The 1 year and 2 year OS and confidence interval will be calculated.
Time Frame: Year 1 and 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
percentage of participants
  1 year | 87.3 [72.1 to 94.5]
  2 years | 82 [65.9 to 91]

2. Secondary Outcome: Relapse/Progression
Description: Relapse is defined as the appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size. Progression is defined as a lymph node with a diameter of the short axis of less than 1.0 cm must increase by >= 50% and to a size of 1.5 x 1.5 cm or more than 1.5 cm in the long axis.
Time Frame: Year 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
percentage of participants | 12.5 [4.5 to 24.8]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: The time to this event is the time from enrollment until death, relapse/progression, receipt of anti-lymphoma therapy, or last follow up, whichever comes first. Progression-free survival (PFS) will be estimated using the Kaplan Meier product limit estimator. The PFS probability and confidence interval will be calculated at two years post-transplant.
Time Frame: Year 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
percentage of participants | 79.8 [63.7 to 89.4]

4. Secondary Outcome: Complete Remission (CR) and/or Partial Response (PR)
Description: The frequencies and proportions of patients who have a CR or PR. CR is defined as the disappearance of all evidence of disease, and PR is defined as the regression of measurable disease and no new sites.
Time Frame: Day 100
Population: One participant died at day 64 and was not included in analysis
Measure: Number; unit: participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 39
participants
  CR | 36
  PR | 1
  Relapse/Progression | 2

5. Secondary Outcome: Time to Progression After CR
Description: This will be assessed in patients with CR. Patients are considered failure for this end point if they relapse after complete remission. Surviving patients with no history of relapse/progression are censored at time of last follow-up.
Time Frame: Year 2
Population: No data collected to analyze this outcome measure
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 0

6. Secondary Outcome: Lymphoma Disease-free Survival
Description: This will be assessed in patients with CR. Patients are considered failure for this end point if they die or if they relapse after complete remission. Patients with no history of relapse or death after complete remission are censored at time of last follow up.
Time Frame: Year 2
Population: No data collected to analyze this outcome measure.
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 0

7. Secondary Outcome: Cumulative Incidence of Neutrophil Recovery
Description: Neutrophil recovery is defined as two consecutive days of absolute neutrophil count (ANC) > 500 neutrophils/μL following the expected nadir.
Time Frame: Day 28
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
percentage of participants | 97.5 [77.7 to 99.7]

8. Secondary Outcome: Cumulative Incidence of Platelet Recovery
Description: Platelet recovery is defined as a platelet count greater than 20,000/μL for the first of two consecutive labs with no platelet transfusions 7 days prior.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
percentage of participants | 92.5 [75.9 to 97.8]

9. Secondary Outcome: Hematologic Function
Description: Hematologic function will be defined as ANC > 1500 neutrophils/μL, Hemoglobin> 10g/dL without transfusion support, and platelets > 100,000/μL
Time Frame: Days 100 and 365
Measure: Number; unit: participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
participants
  Day 100 | 11
  Day 365 | 23

10. Secondary Outcome: Number of Participants Experiencing Toxicity
Description: Toxicities will be defined by using the version 3.0 NCI Common Terminology Criteria for Adverse Events (CTCAE) criteria. Only grade 3 and higher toxicities will be collected.
Time Frame: Year 2
Measure: Number; unit: participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
participants | 9

11. Secondary Outcome: Number of Participants Experiencing Infections
Description: Microbiologically documented infections will be reported by site of disease, date of onset, severity, and resolution, if any.
Time Frame: Year 1
Measure: Number; unit: participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
participants | 22

12. Secondary Outcome: Treatment-Related Mortality (TRM)
Description: TRM is defined as death occurring in a patient from causes other than relapse or progression. A cumulative incidence curve will be computed along with a 95% confidence interval at 100 days post-transplant.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
percentage of participants | 5.2 [0.9 to 15.2]

13. Secondary Outcome: Immunologic Reconstitution
Description: Immunologic Reconstitution will be assessed by quantitative immunoglobulin measurement (IgM, IgG and IgA)
Time Frame: Year 1
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 40
mg/dL
  IgG | 1090 [270 to 2331]
  IgA | 123 [6 to 534]
  IgM | 48.5 [24 to 254]

14. Secondary Outcome: HIV Single-Copy Polymerase Chain Reaction (PCR)
Description: HIV RNA assay will be performed at the specified time points and summarize the assessments of the viral copy number using descriptive statistics.
Time Frame: Baseline, Days 100, 180, 365, and 730
Population: Participants with an undetectable (<50 copies/mL) viral load are not included in this analysis (Baseline = 32, Day 100 = 19, Day 180 = 20, Day 365 = 19, and Day 730 = 21)
Measure: Median (Full Range); unit: copies/mL
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 32
copies/mL
  Baseline | 80 [50 to 17455]
  Day 100 | 298 [58 to 1100]
  Day 180 | 84 [55 to 36815]
  Day 365 | 97 [75 to 5097]
  Day 730 | 130 [75 to 351]

15. Secondary Outcome: Microbial Translocation Markers
Description: Level of microbial translocation markers will be determined by nonparametric Mann-Whitney tests comparing the distribution of prior microbial translocation markers between patients.
Time Frame: Day 30 and 100
Population: No data collected to analyze this outcome measure.
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 0

16. Secondary Outcome: Ig and Epstein-Barr Virus (EBV) DNA in Blood
Description: The presence of clonal Ig DNA in plasma will be assessed, as will EBV copy number in plasma and in peripheral blood
Time Frame: Day 100, 180, and 365
Population: No data collected to analyze this outcome measure.
Arm/Group | Autologous Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years post-transplant
Description: Serious Adverse Events (AE) are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected grades 3-5 adverse events were required to be reported through the AE system per protocol.
Arm/Group | Autologous Transplant
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 3/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Transplant (N=40)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Transplant (N=40)
Appendicitis (Infections and infestations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2010-04-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT01141712/Prot_SAP_ICF_000.pdf